CLINICAL TRIAL: NCT02212587
Title: Pilot Study of the in Vivo Efficacy of Tobramycin Inhalation Powder (TIP) in Cystic Fibrosis Patients Infected With Burkholderia Cepacia Complex
Brief Title: Tobramycin Inhalation Powder (TIP) in Cystic Fibrosis Patients Infected With Burkholderia Cepacia Complex
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TIPBCC002; 165476 (Other: Health Canada)
Record Dates: First submitted 2014-08-06; First posted 2014-08-08 (Estimated); Results first posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Cystic Fibrosis; Burkholderia Cepacia Infection
Keywords: inhaled antibiotics
MeSH Terms: conditions — Cystic Fibrosis; Burkholderia Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TOBI Podhaler (Experimental)
  Interventions: Drug: TOBI

INTERVENTIONS:
Drug: TOBI — New inhalation devices such as the podhaler can administer tobramycin inhalation powder TIP/TOBI and achieve very high sputum drug levels. TOBI will be administered using the Podhaler

SUMMARY:
The objective of this study is to determine if tobramycin inhalation powder (TIP) can reduce the amount of Burkholderia Cepacia Complex (BCC) species - type of bacteria, in the sputum of cystic fibrosis patient.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 years or older
* Diagnosis of CF based on the following: sweat chloride>60 mEq/L or genotype with 2 identifiable mutations consistent with CF; and one or more clinical features consistent with CF.
* Chronically infected with a Burkholderia cepacia complex species (>50% of respiratory specimens positive in the 24 months prior to screening).
* Able to produce sputum (expectorated or induced).
* Able to reproducibly perform pulmonary function testing.
* Written informed consent provided.

Exclusion Criteria:

* Post lung transplantation.
* Pregnancy.
* Acute exacerbation requiring IV or oral antibiotics within 14 days
* Patients currently receiving inhaled tobramycin/TOBI
* A septic or clinically unstable patient, as determined by the investigator.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Waters, MD, Principal Investigator — Hospital of Sick Children
Locations (2):
- Canada (2):
  - St. Michael's Hospital, Toronto, Ontario
  - Hospital for Sick Children, Toronto, Ontario

REFERENCES:
- [Result] Waters V, Yau Y, Beaudoin T, Wettlaufer J, Tom SK, McDonald N, Rizvi L, Klingel M, Ratjen F, Tullis E. Pilot trial of tobramycin inhalation powder in cystic fibrosis patients with chronic Burkholderia cepacia complex infection. J Cyst Fibros. 2017 Jul;16(4):492-495. doi: 10.1016/j.jcf.2017.02.008. Epub 2017 Mar 3. PMID 28262569

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TOBI Podhaler
Started | 10
Completed | 9
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | TOBI Podhaler
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Region of Enrollment [Number; unit: participants]
  Canada | 10
Burkholderia cenocepacia IIIA, n (%) [Count of Participants; unit: Participants] | 4
Burkholderia cenocepacia IIIB, n (%) [Count of Participants; unit: Participants] | 3
Burkholderia multivorans, n (%) [Count of Participants; unit: Participants] | 3
Sputum density log10 CFU/ml, median (range) [Median (Full Range); unit: log10 CFU/ml] | 7.9 [3.1 to 8.8]

OUTCOME MEASURES:

1. Primary Outcome: The Change in Sputum Density of BCC in Colony Forming Units (CFUs)/ml From Day 0 to Day 28 of TIP Treatment.
Description: The change in sputum density of BCC in colony forming units (CFUs)/ml from day 0 to day 28 of TIP treatment. Sputum density was calculated by doing serial dilutions of sputum on agar plates and counting colony forming units expressed per ml.
Time Frame: 0 to 28 days
Population: sputum density measurements was calculated for all patients from Day 0 to Day 28
Measure: Mean (Full Range); unit: CFU/ml log10
Arm/Group | TOBI Podhaler
Number analyzed (Participants) | 10
CFU/ml log10 | -1.4 [-3.9 to 0.8]

2. Secondary Outcome: The Change in Pulmonary Function Tests, Including Forced Expiratory Volume in 1 Second (FEV1), Forced Vital Capacity (FVC) and Maximal Mid-expiratory Flow Rate (FEF25-75), Measured at Day 0 and Day 28 of TIP Treatment.
Description: The main lung function measure was relative change in FEV1 from day 0 to Day 28 reported as %.
Time Frame: 0 to 28 days
Population: All patients had lung function measures which were analyzed.
Measure: Mean (Full Range); unit: relative change in FEV1 expressed as %
Arm/Group | TOBI Podhaler
Number analyzed (Participants) | 10
relative change in FEV1 expressed as % | 4.6 [-6.6 to 28.1]

3. Other Pre Specified Outcome: The Change in the Measurement of Markers of Pulmonary Inflammation (Neutrophil Counts, Neutrophil Elastase and IL-8 Levels in Sputum) Measured at Day 0 and Day 28 of TIP Treatment.
Description: We measured both neutrophil elastase sputum for participants.
Time Frame: 0 to 28 days
Population: Sputum inflammatory markers were measured for 8 participants who could produce sputum.
Measure: Mean (Full Range); unit: NE = ug/ml
Arm/Group | TOBI Podhaler
Number analyzed (Participants) | 8
NE = ug/ml | -51.9 [-188.4 to 47.3]

4. Other Pre Specified Outcome: Trough and Peak Sputum Tobramycin Concentration Measured on Day 28 of TIP Treatment.
Description: We did trough (0 hour) and peak (1 hour post dose) TIP sputum tobramycin concentrations and reported it for participants.
Time Frame: Day 28
Population: We did pre and post TIP sputum tobramycin concentrations in 9 participants at Day 28 since one patient stopped taking the drug.
Measure: Median (Full Range); unit: ug/ml
Arm/Group | TOBI Podhaler
Number analyzed (Participants) | 9
ug/ml
  Trough (0 hr) | 194 [11 to 2100]
  Peak (1 hr post dose) | 1025 [306 to 4700]

5. Other Pre Specified Outcome: The Change in BCC Planktonic and Biofilm MICs to Tobramycin Measured on Day 0 and on Day 28 of TIP Treatment.
Description: For all participants, the minimum inhibitory concentration of tobramycin for planktonic and biofilm grown BCC was measured in the lab on the isolate collected before and after TIP treatment.
Time Frame: 0 to 28 days
Measure: Mean (Full Range); unit: ug/ml (MIC50)
Arm/Group | TOBI Podhaler
Number analyzed (Participants) | 10
ug/ml (MIC50)
  Day 0 | 200 [10 to 1600]
  Day 28 | 400 [10 to 1600]

6. Other Pre Specified Outcome: The Number of Participants With Adverse Events Measured at Day 14 and at Day 28 of TIP Treatment.
Description: The number of participants with adverse events was reported for all participants in the trial.
Time Frame: At Dat 0, Day 14, and Day 28
Population: We observed for adverse events in all participants and reported on those that had an adverse event.
Measure: Count of Participants; unit: Participants
Arm/Group | TOBI Podhaler
Number analyzed (Participants) | 10
Participants | 6

7. Other Pre Specified Outcome: The Change in the Measurement of Markers of Pulmonary Inflammation (Neutrophil Counts, Neutrophil Elastase and IL-8 Levels in Sputum) Measured at Day 0 and Day 28 of TIP Treatment.
Description: We measured both IL-8 sputum for participants.
Time Frame: 0 to 28 days
Population: Sputum inflammatory markers were measured for 8 participants who could produce sputum.
Measure: Mean (Full Range); unit: IL-8 = ng/ml
Arm/Group | TOBI Podhaler
Number analyzed (Participants) | 8
IL-8 = ng/ml | -127 [-298.62 to 101.8]

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | TOBI Podhaler
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No